CLINICAL TRIAL: NCT00051714
Title: Early Primary Prevention of Conduct Problems
Brief Title: Early Prevention of Conduct Problems
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Laurie Brotman, Professor Science Professor of Child & Adolescent Psychiatry, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH055188 (NIH); R01MH055188 (NIH); DSIR 84-CTP
Record Dates: First submitted 2003-01-15; First posted 2003-06-04 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Conduct Disorder
Keywords: Social Behavior Disorders
MeSH Terms: conditions — Conduct Disorder

ARMS (1):
- Early Primary Prevention (Experimental)
  Interventions: Behavioral: Family-Based Preventive Intervention

INTERVENTIONS:
Behavioral: Family-Based Preventive Intervention

SUMMARY:
The purpose of this study is to examine the immediate and long-term effects of a prevention program in children at risk for developing conduct problems and antisocial behavior.

DETAILED DESCRIPTION:
Participants are randomly assigned to a year-long family-based intervention or to a no contact control group. The intervention focuses on improving parenting practices, parent-child interactions, and child social competence.

Children are assessed at the beginning of the study and again after one year. The development of conduct problems, social competence, and school functioning is assessed from second through fifth grade. Assessments are made through observations, parent and teacher ratings, and diagnostic interviews.

ELIGIBILITY:
Inclusion Criteria:

* Sibling of youth adjudicated in Family Court

Ages: 33 Months to 63 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1050 (Actual)
Dates: Start 1997-03; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
behavior problems | March 1997 - December 2012

CONTACTS AND LOCATIONS:
Locations (1):
- New York University Child Study Center, New York, New York, United States